CLINICAL TRIAL: NCT07323719
Title: Comparison Between Topical N-acetyl Cysteine (NAC) in Cold Cream Versus Cold Cream in Mild and Moderate Atopic Dermatitis: Clinical and Bacteriological Evaluation. A Randomized Control Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar Saeed Salim, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-224-2024
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (AD)
Keywords: N-acetyl cystiene, Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- n-acetyl cyteine arm (Experimental): the interventional arm recieves n-acetyl cyteien 10% in cold cream twice daily on the lesion
  Interventions: Drug: n-acetyl cyteien
- control arm (Placebo Comparator): recieve cold cream twice daily on affected lesion
  Interventions: Drug: cold cream

INTERVENTIONS:
Drug: n-acetyl cyteien — n-acetyl cyteien 10% in cold cream
  Arms: n-acetyl cyteine arm
Drug: cold cream — cold cream is made of vaseline ,bees wax and other emollients as a placebo arm
  Arms: control arm

SUMMARY:
Atopic dermatitis (AD), or atopic eczema, is a chronic relapsing, inflammatory skin disease, characterized by intense pruritus that leads to considerable burden on patients' quality of life (Sidbury et al., 2023). The dramatic rise of AD prevalence in the past half century is well documented, with prevalence reaching 15-30% of children and 2-10% of adults worldwide. Onset of the disease usually starts in childhood and although most cases resolve by adolescence, a fraction remains afflicted in adulthoodThe exact etiopathogenisis of AD is not well understood, being a complex interplay between genetic, environmental and immunological factors (Serra-Baldrich et al., 2017). Cutaneous flora imbalance in AD is well established. In particular, Staph aureus colonization is found in the vast majority of AD patients, especially in the sweat gland ducts (Gonzalez et al., 2017). Some studies found that the prevalence of Staph aureus colonization exceeds 90% of AD patients in comparison to most healthy people. In Staph. aureus- colonized AD patients, the Staph. aureus density in lesional skin was found to be more than in non-lesional skin. Recently, a temporal relationship between Staph. aureus density and clinical severity of AD was found, strongly implicating Staph. aureus in disease pathogenesis (Di Domenico et al., 2019; Ogonowska et al., 2021). Atopic dermatitis-derived Staphylococcus. epidermidis strains elicit higher inflammatory response than healthy strains.it was found that Staph. epidermidis in AD triggers inflammation by activating NF-kappa B, induces pro-inflammatory cytokines, downregulates skin barrier molecules like filaggrin and it is more prevalent in severe cases(Ochlich et al., 2023). After antimicrobial therapies targeting reduction of Staphylococcus colonization, clinical symptoms significantly decline along with resettling of diverse microflora (Brüssow, 2016). However, the propensity of Staph. aureus and Staph. epidermidis to form protective biofilms and rapid emergence of antibiotic resistance pose grave concern and prompt the search for other antimicrobial agents with less risk of resistance such as non-antibiotic antimicrobial agents and phototherapy (Brockow et al., 1999; Gonzalez et al., 2017; Man et al., 2017). Despite advances in systemic therapy for AD, topical therapies remain the mainstay of treatment due to their proven efficacy to alleviate inflammation and pruritus and generally favorable safety profile. They include emollients,corticosteroids, calcineurin inhibitors and antimicrobials (Sidbury et al., 2023).

N-acetyl cysteine (NAC) is a widely used drug in human clinical practices. It has been systemically used in the treatment of acetaminophen toxicity and as a mucolytic agent in the treatment of lower respiratory tract diseases, and its uses is recently increasing. (Janeczek et al., 2019). Regarding dermatological applications; Efficacy of N-acetyl cysteine was shown in excoriation disorder, onychophagia disorder, trichotillomania, acne vulgaris, Type I lamellar ichthyosis, bullous morphea, systemic sclerosis, toxic epidermal necrolysis, atopic dermatitis, xeroderma pigmentosum, and pseudoporphyria. Studies also show benefits in wound healing and photoprotection (Janeczek et al., 2019). N-acetyl cysteine also has antioxidant, cytoprotective, anti-inflammatory and antimicrobial properties. Oxidative stress contributes to barrier dysfunction in AD. NAC is a precursor of glutathione, a potent antioxidant which improves the barrier function. NAC also modulates cytokine production: tumor necrosis factor-alpha (TNF-α) and interleukins (IL-6 and IL-1β) by suppressing the activity of nuclear factor kappa B (NF-κB), potentially reducing the inflammatory response associated with Staph. aureus colonization. (Tenório et al., 2021) In addition, the published literature shows that NAC has an adverse effect on biofilm formation and impedes its formation at various stages. N-acetyl cysteine, as an acidic compound, applied at high concentrations, was able to penetrate the biofilm and bacterial membrane and increase the intracellular oxidative status and halt protein synthesis, in this way killing the bacterial cells (Li et al., 2020).Regarding skin hydration; NAC solution (20 w/v%) was applied to the forearm skin twice a day for 4 weeks resulted in increased skin hydration in 9/11 AD patients and decreased TEWL in 9/10 AD patients (Nakai et al., 2015). N-acetyl cysteine restored the expression of some cell adhesion molecules that contribute to forming the skin barrier in a mouse model of AD by reducing oxidative stress. Therefore, the topical application of NAC may have increased skin hydration and decreased Trans-epidermal water loss (TEWL) by strengthening the function of this barrier (Nakai et al., 2017).

DETAILED DESCRIPTION:
Despite NAC relevant therapeutic potential, in several experimental studies, its effectiveness in clinical trials, addressing different pathological conditions, is still limited. Only one cohort study was done on humans using 20% NAC solution but 10% NAC in cold cream was the maximum concentration feasible for manufacture for our study. We first conducted a pilot study on 7 patients and it showed clinical improvement together with reduction in the colony count of Staph. aureus, therefore we decided to test this concentration on a larger scale. To the best of our knowledge, this is the first RCT conducted on atopic dermatitis patients using 10% NAC in cold cream.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atopic dermatitis defined according to Hanifin and Rajka criteria, with mild to moderate degree according to EASI score

Exclusion Criteria:

* -Severe or erythrodermic patients and those indicated for more aggressive systemic immune suppressive therapy.
* Patients with oozing or infected lesions
* Patients receiving systemic treatment within one month or topical treatment within 2 weeks before enrollment into the study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
microbial improvement | 4 weeks from starting treatment
  - Percentage of reduction of Staphylococcus aureus and Staphylococcus epidermidis load on the skin of treated patients at EOT or EOS whichever earlier, as assessed quantitatively by Colony Forming Units (CFU) and comparing percentage of reduction between the two groups.
clinical improvement | 4 weeks from starting treatment
  - Percentage of clinical improvement using local EASI score for the chosen lesion at EOT (70% improvement or more) and comparing percentage of clinical improvement between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Samar Ragaie El-tahlawi, Professo, Study Director — Cairo University
Locations (1):
- Cairo Unversity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
i would ask for participants permission first